CLINICAL TRIAL: NCT03538912
Title: Impact of the Use of Biomarkers on Early Discontinuation of Empirical Antifungal Therapy in Critically Ill Patients: a Randomized Controlled Study.
Brief Title: Early Discontinuation of Empirical Antifungal Therapy and Biomarkers
Acronym: SEAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017_07; 2017-003793-13 (EudraCT Number)
Record Dates: First submitted 2018-04-25; First posted 2018-05-29 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Invasive Candidiasis
Keywords: empirical antifungal therapy; invasive candidiasis; biomarkers; de-escalation; ICU
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biomarker group (Other): patient follow the Biomarker strategy
  Interventions: Other: Biomarker strategy
- Routine group (Other): patient follow the routine strategy
  Interventions: Other: Routine strategy

INTERVENTIONS:
Other: Biomarker strategy — EAT duration is determined by β-D-1,3-glucan and mannan serum assays, performed at day 0 (day of EAT initiation) and day 3.
  Arms: Biomarker group
Other: Routine strategy — EAT duration is based on IDSA guidelines, which recommend 14 days of treatment for patients without subsequent proven ICI, and who improve under antifungal treatment, or less in other situations.
  Arms: Routine group

SUMMARY:
Empirical antifungal therapy (EAT) is frequently prescribed to septic critically ill patients with risk factors for invasive Candida infections (ICI). However, among patients without subsequent proven ICI, antifungal discontinuation is rarely performed, resulting in unnecessary antifungal overuse.

The investigators postulate that the use of fungal biomarkers could increase the percentage of early discontinuation of EAT among critically ill patients suspected of ICI, as compared with a standard strategy, without negative impact on day 28-mortality.

To test this hypothesis, the investigators designed a randomized controlled open-label parallel-group study.

DETAILED DESCRIPTION:
Patients requiring EAT will be randomly assigned to:

* intervention group: a strategy in which EAT duration is determined by (1,3)-B-Dglucan and mannan serum assays, performed on day 0 (day of EAT initiation) and day 3. Early stop recommendation, provided before day 7, will be determined using an algorithm based on the results of biomarkers.
* control group: a routine care strategy, based on international guidelines, which recommend 14 days of treatment for patients without subsequent proven ICI, and who improve under antifungal treatment, or less in other situations.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years
* Who require EAT for the first time in the ICU (this treatment is prescribed based on the presence of risk factors and clinical suspicion of ICI)
* With an expected ICU length of stay of at least 6 days after EAT initiation
* Informed written consent

Exclusion Criteria:

* Neutropenia (neutrophil count <500 cells /µL)
* Active malignant hemopathy
* Bone marrow transplantation in the last 6 months
* Polyvalent immunoglobulins in the past months
* Documented ICI in the past 3 months
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
percentage of patients receiving early discontinuation of EAT, defined as a discontinuation strictly before day 7 after EAT initiation | day 7 after EAT initiation
  This trial is designed to demonstrate whether, in critically ill patients suspected for ICI, the biomarker strategy, as compared with a standard strategy, is at the same time:
  1. superior in terms of antifungal use and
  2. Non-inferior in terms of death

SECONDARY OUTCOMES:
death from any cause | day 28 after EAT initiation
  This trial is designed to demonstrate whether, in critically ill patients suspected for ICI, the biomarker strategy, as compared with a standard strategy, is at the same time:
  1. superior in terms of antifungal use and
  2. Non-inferior in terms of death
percentage of patients who presented a proven ICI after EAT discontinuation | at day 28 or ICU discharge, if it occurs before day 28
percentage of patients who received at least two periods of antifungal treatment (prescribed for separate episodes of suspected or proven ICI) | at day 28 or ICU discharge, if it occurs before day 28
intensity of Candida colonization during ICU stay | at day 28 or ICU discharge, if it occurs before day 28
  Five body sites (among urine, anal swabs, pharyngeal swabs, nasal swabs, axillary swabs, gastric aspirates if patients have a nasogastric tube, and tracheal aspirates if patients are intubated or have a tracheotomy) are sampled on day 0 and then once per week for the semi-quantitative determination of yeast colonisation. The number of colony-forming units is scored as follows: score 1, <10 colony-forming units; score 2, 10 to 50 colony-forming units; score 3, >50 colony-forming units; score 4, >50 colony-forming units confluent. Intensity of colonization is determined for each date of sampling, by dividing the sum score for each colonized site by the number of sites sampled giving a mean Candida load. An overall score of >4 is possible in the case of isolation of several Candida species.
percentage of patients colonized with a resistant strain of Candida | at day 28 or ICU discharge, if it occurs before day 28
antifungal-free days | at day 28 or ICU discharge, if it occurs before day 28
ventilator-free days | at day 28 or ICU discharge, if it occurs before day 28
ICU-free days | at day 28 or ICU discharge, if it occurs before day 28
ICU mortality | at day 28 or ICU discharge, if it occurs before day 28
day 90 mortality | at day 90
Characterization of the fungal intestinal microbiota studied by standard mycology | at baseline, at Day 7, day 14 day 21 and day 28
Characterization of the fungal intestinal microbiota studied by metagenomics | at baseline, at Day 7, day 14 day 21 and day 28
Characterization of the bacterial intestinal microbiota studied by culture bacteriology | at baseline, at Day 7, day 14 day 21 and day 28

CONTACTS AND LOCATIONS:
Overall Officials: Anahita Rouze, MD, Principal Investigator — University Hospital, Lille
Locations (10):
- France (10):
  - CH ARRAS, Arras
  - CH de DOUAI, Douai
  - CH Dunkerque, Dunkirk
  - Centre Hospitalier Dr Schaffner, Lens
  - Ch Dr.Schaffner de Lens, Lens
  - Hôpital Roger Salengro, CHU, Lille
  - CH Roubaix, Roubaix
  - CHU de Rouen, Rouen
  - Ch Tourcoing, Tourcoing
  - Centre hospitalier de valenciennes, Valenciennes